CLINICAL TRIAL: NCT00188045
Title: Hemodynamic Effects of Chronic Administration of Spironolactone, Propranolol and Their Association in Alcoholic Cirrhotic Patients
Brief Title: Hemodynamic Effects of Chronic Administration of Spironolactone and/or Propranolol in Alcoholic Cirrhotic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHRC 01-13
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2001-12

CONDITIONS: Alcoholic Cirrhosis
Keywords: Portal hypertension, alcoholic cirrhosis, Hepatic venous pressure gradient, hemodynamic, spironolactone, propranolol
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Hypertension, Portal

INTERVENTIONS:
Drug: Propranolol - Spironolactone

SUMMARY:
The aim of this study was assesment of splanchnic and systemic hemodynamic effects of chronic administration (2 month) of spironolactone or propranolol, alone or in association in alcoholic cirrhotic patients. The patients were randomized in 4 groups (aldactone 150 mg/day, propranolol 160 mg/day, aldactone 150 mg/day + propranolol 160 mg/day, placebo). Systemic and splanchnic hemodynamic effect were evaluated by hepatic venous pressure gradient measurements before and after 2 month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Indication of transjugular hepatic biopsy
* alcoholic cirrhosis
* presence of oesophageal varices ≤ stade 2

Exclusion Criteria:

* renal insufficiency
* natremia ≤ 135 mmol/l
* vasoactive treatment in the last month before inclusion
* hepatocellular carcinoma
* positive HIV and HCV patients
* paracentesis in the last week before inclusion
* digestive bleeding in one last week
* oesophageal varices stade 3 or 2 with red signs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 1995-04; Study Completion 2003-12

PRIMARY OUTCOMES:
assessment of hepatic veinous pressure gradient changes after chronic treatment by spironolactone or propranolol alone or in association.

SECONDARY OUTCOMES:
Efficacy of spironolactone/propranolol association

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cales, PHD, Principal Investigator — UH Angers